CLINICAL TRIAL: NCT02001662
Title: The Analgesic Efficacy of the Adductor Canal Blockade in High Pain Responders After Arthroscopic Knee Surgery - a Randomized Clinical Trial
Brief Title: Adductor Canal Block and Arthroscopic Knee Surgery, High Pain Responders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Malene Espelund, MD,, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM3-ME-13; 2013-000663-83 (EudraCT Number); H-3-2013-039 (Other: Regional Ethics Committee, Capital region of Denmark)
Record Dates: First submitted 2013-04-09; First posted 2013-12-05 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-12

CONDITIONS: Arthroscopic Knee Surgery
Keywords: Minor arthroscopic knee surgery including ACL-reconstruction (hamstrins graft); High pain responders; Adductore Canal Block; Analgesics; Ultrasound guided nerve block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group, block no. 1 - Ropivacain (Experimental): Adductor-Canal-Block no.1: 30mL ropivacaine (7.5 mg/ml) when postoperative VAS-score is > 40mm (on a 0-100 mm VAS-scale) during a 45 degree active flexion of the knee.
  Adductor-Canal-Block no.2: after 45 min (t45) - 30mL isotonic saline.
  Interventions: Procedure: Intervention group, block no. 1 - Ropivacain
- Control group, block no. 1 - saline (Sham Comparator): Adductor-Canal-Block no.1: 30mL isotonic saline when postoperative VAS-score is above 40mm (on a 0-100 mm VAS-scale) during a 45 degree active flexion of the knee.
  Adductor-Canal-Block no.2: after 45 min (t45) - 30mL ropivacaine (7.5 mg/ml)
  Interventions: Procedure: Control group: 1. block - saline

INTERVENTIONS:
Procedure: Intervention group, block no. 1 - Ropivacain — Intervention group: 1. block ropivacaine - 2. block saline
  Arms: Intervention group, block no. 1 - Ropivacain
Procedure: Control group: 1. block - saline — Control group: 1. block saline - 2. block ropivacaine
  Arms: Control group, block no. 1 - saline

SUMMARY:
The investigators want to explore the analgesic effect of Adductor Canal Blockade (a peripheral nerve block) in high pain responding patients after arthroscopic knee surgery. The investigators hypothesize that the nerve block will have an abrupt analgesic effect.

ELIGIBILITY:
Inclusion Criteria:

Arthroscopic knee surgery, if reconstruction of Anterior Cruciate Ligament only hamstring graft 18-80 years of age BMI 18-40 ASA I-III written Consent

Exclusion Criteria:

Unable to communicate in danish, allergic reactions toward any study medication pregnancy alcohol/drug abuse daily opioid consumption scin infection (injection site)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Pain score during 45 degree flexion of the knee | 45 minutes after nerve block
  Pain score during flexion of the knee 45 min. after nerve block

SECONDARY OUTCOMES:
Pain score | 0-90 min. after first nerveblock
  pain score at rest: time 0,15,30,45,60,75,90 min. after first nerve block pain score during flexion of the knee: time 0,15,30,45,60,75,90 min. after first nerve block pain score during mobilisation (5m walk): 45 and 90 min after nerve block
muscle strength | 45 and 90 min after nerve block
  patients accesses muscle strength during walk
Opioid consumption | 0-90 min after nerve block

CONTACTS AND LOCATIONS:
Overall Officials: Malene Espelund, MD, Principal Investigator — Glostrup University Hospital, University of Copenhagen
Locations (1):
- Amager Hospital, University of Copenhagen, Denmark, Copenhagen, Copenhagen, Amager, Denmark